CLINICAL TRIAL: NCT06361576
Title: Patients With Upper Gastrointestinal Adenocarcinoma Enrolled in a Patient Support Program to Receive Nivolumab in the Metastatic Setting: Real-World Data From Canada
Brief Title: Real-World Use of Nivolumab for the Treatment of Patients With Metastatic Upper Gastrointestinal Cancer in Canada
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-1443
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Upper Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants enrolled and treated with nivolumab in the metastatic setting
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — As per product label

SUMMARY:
The purpose of this observational study is to describe the demographics, and disease characteristics of participants with metastatic upper gastrointestinal cancer, along with the treatment characteristics of these patients when treated with nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Bristol-Myers Squibb GastroEsophageal Opdivo in non-Resectable, advanced or metastatic Adenocarcinoma Patient Support Program (GEORgiA PsP) in Canada
* Have consented to the use of their de-identified data generated from information collected during the course of the GEORgiA PsP

Exclusion Criteria:

* Aged <18 years
* HER2 positive status
* Untreated brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of individuals diagnosed with HER2 negative, unresectable, advanced or metastatic gastric cancer, gastroesophageal junction cancer or esophageal adenocarcinoma (GC/GEJC/EAC) that participated in the Bristol-Myers Squibb Patient Support Program (PSP) in Canada, GEORgiA PSP (GastroEsophageal Opdivo in non-Resectable, advanced or metastatic Adenocarcinoma)
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Particpant sociodemographics | Baseline
Participant Eastern Cooperative Oncology Group (ECOG) score | Baseline
Participant HER2 status | Baseline
Participant comorbidities | Baseline
Participant tumour location | Baseline
Participant treatment history | Baseline

SECONDARY OUTCOMES:
Initial nivolumab dosage prescribed to participants | Index date
Number of nivolumab treatments received by participants | Up to 75 weeks
Planned combination chemotherapy treatment | Index date
Nivolumab treatment initiation date | Index date
Nivolumab dosage modification | Up to 75 weeks
Participant treatment duration | Up to 75 weeks
Reason for participant discharge | Up to 75 weeks
Participant adverse events (AEs) | Up to 75 weeks
Management of participant adverse events (AEs) | Up to 75 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bayshore Specialty Rx Ltd., Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts